CLINICAL TRIAL: NCT03261791
Title: A Exploratory Study of Apatinib Adjuvant Therapy for Hepatocellular Carcinoma With Portal Vein Invasion Who Underwent Radical Resection
Brief Title: Adjuvant Therapy With Apatinib for HCC Patients With PVTT Who Underwent Radical Resection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APA- ZS-PVTT
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Carcinoma, Hepatocellular
Keywords: hepatocellular carcinoma; apatinib; portal vein invasion; adjuvant therapy; resection
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib (Experimental): Apatinib mesylate tablets 500 mg po qd.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib mesylate tablets 500 mg po qd.

SUMMARY:
In this phase 2 study, we aim to evaluate the effects and safety of adjuvant apatinib therapy for the patients who underwent R0 resection for hepatocellular carcinoma with portal vein tumor thrombus.

DETAILED DESCRIPTION:
Portal vein tumor thrombus (PVTT) is one of the characteristics of advanced stage for patients with hepatocellular carcinoma (HCC). There's limited treatment choice for these patients. Even for those who underwent curative resection (R0 resection), the recurrence rate was extremely high. Apatinib is a highly selective VEGFR2 inhibitor and reduces the angiogenesis of tumor efficiently, which had been proven effective in many solid tumors, is a Chinese domestic TKI targeting vascular endothelial growth factor receptor. Phase 2 study of apatinib for patients with advanced HCC had shown signals of clinical efficacy and modest safety. In this study, we aim to evaluate the effects and safety of adjuvant apatinib therapy for the patients who underwent R0 resection for HCC with PVTT.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 18-70 years.
2. HCC diagnosis confirmed by pathological examination who did not receive anti-tumor treatment (anti-tumor treatment including but not limited to: local ablation therapy, TACE, radiation therapy, chemotherapy, targeted drug therapy, etc.)
3. Underwent radical resection for hepatocellular carcinoma with portal vein tumor thrombus, as assessed by preoperative imaging or intraoperative findings, within 4 weeks
4. Child-Pugh class: A or B7
5. The ECOG: 0-1 points
6. The expected survival time ≥ 6 months.
7. Main organs function is normal including:

   * blood routine examination

     * HB ≥ 90 g/L
     * ANC ≥ 1.5×109 /L
     * PLT ≥ 80×109/L
   * biochemical test

     * ALB ≥ 29 g/L
     * ALT<3 ULN and AST< 3 ULN
     * TBIL ≤ 1.5 ULN
     * Serum creatinine ≤ 1.5 ULN；
8. Women of childbearing age must have pregnancy tests (serum or urine) within 7 days prior to admission, and the results are negative and are willing to use appropriate methods of contraception at 8 weeks after the trial and at the end of the test. For men, surgical sterilization should be applied, or consent to the appropriate method of contraception 8 weeks after the trial and at the end of the trial;
9. subjects voluntarily joined the study, signed informed consent, good compliance, and followed up.

Exclusion Criteria:

1. Hepatic duct carcinoma、mixed cell carcinoma and fiberboard layer cell carcinoma which have confirmed; Past (5 years) or current with other malignant tumor, except skin basal cell carcinoma and cervical carcinoma in situ.
2. Patients with hypertension who are unable to fall within normal range by antihypertensive medications (systolic pressure > 140 mmHg, diastolic pressure > 90 mmHg).
3. With the second level of myocardial ischemia or myocardial infarction, poor control of the arrhythmia (including QTc interval = 450 ms, male female = 470 ms).
4. Factors that affect oral medication, such as inability to swallow, chronic diarrhea and intestinal obstruction, which significantly affect the use and absorption of drugs.
5. Ascites with clinical symptoms requires therapeutic peritoneal paracentesis or drainage.
6. In the past 6 months, with the history of alimentary tract hemorrhage or definite gastrointestinal bleeding tendency, such as: the risk of bleeding esophageal varices, local active ulcerative lesions, fecal occult blood; For those with fecal occult blood (+), gastroscopy is required.
7. Abdominal fistula, gastrointestinal perforation, or abdominal abscess occurred within 28 days before entry;
8. Postoperative complications were not relieved.
9. Abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN+4 seconds), with bleeding tendency or undergoing thrombolysis or anticoagulant therapy;
10. Past and present pulmonary fibrosis history, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug associated pneumonia, and severe lung function impairment;
11. Urine routine showed that urinary protein is more than + + or confirmed 24 hours urine protein is more than 1.0 g;
12. Symptomatic metastasis of the central nervous system;
13. Pregnant or lactating women; fertile patients who are unwilling or unable to adopt effective contraceptives;
14. Patient with mental illness or a history of psychotropic substance abuse;
15. HIV infection;
16. Before operation, AFP or PIVKA-2 increased, but not decreased to normal range;
17. HBV-DNA>10^3 copys/ml；
18. Other conditions that the investigators considered that not unsuitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2020-01-20 (Estimated); Study Completion 2020-04-20 (Estimated)

PRIMARY OUTCOMES:
recurrence-free survival | 24 months
  From the date of liver surgery to the date of diagnosis of tumor recurrence

SECONDARY OUTCOMES:
overall survival | 24 months
  From the date of liver surgery to the date of death
safety: the potential side effects | 24 months
  The potential side effects

CONTACTS AND LOCATIONS:
Overall Officials: Hui-CHuan Sun, MD&PhD, Principal Investigator — Fudan University; Jia Fan, MD&PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang ZM, Lai EC, Zhang C, Yu HW, Liu Z, Wan BJ, Liu LM, Tian ZH, Deng H, Sun QH, Chen XP. The strategies for treating primary hepatocellular carcinoma with portal vein tumor thrombus. Int J Surg. 2015 Aug;20:8-16. doi: 10.1016/j.ijsu.2015.05.009. Epub 2015 May 27. PMID 26026424
- [Background] Omata M, Lesmana LA, Tateishi R, Chen PJ, Lin SM, Yoshida H, Kudo M, Lee JM, Choi BI, Poon RT, Shiina S, Cheng AL, Jia JD, Obi S, Han KH, Jafri W, Chow P, Lim SG, Chawla YK, Budihusodo U, Gani RA, Lesmana CR, Putranto TA, Liaw YF, Sarin SK. Asian Pacific Association for the Study of the Liver consensus recommendations on hepatocellular carcinoma. Hepatol Int. 2010 Mar 18;4(2):439-74. doi: 10.1007/s12072-010-9165-7. PMID 20827404
- [Derived] Sun HC, Zhu XD, Zhou J, Gao Q, Shi YH, Ding ZB, Huang C, Qiu SJ, Ren N, Shi GM, Sun J, Ye QH, Huang XW, Yang XR, Fan J. Adjuvant apatinib treatment after resection of hepatocellular carcinoma with portal vein tumor thrombosis: a phase II trial. Ann Transl Med. 2020 Oct;8(20):1301. doi: 10.21037/atm-20-6181. PMID 33209881
- See also: Apatinib in Chinese patients with advanced hepatocellular carcinoma: A phase II randomized, open-label trial — http://ascopubs.org/doi/abs/10.1200/jco.2014.32.15_suppl.4019